# **Evaluation of the Efficacy of Different Drugs in the Treatment of Pain in Patients with Temporomandibular Disorder**

Levent Ciğerim DDS, PhD <sup>1</sup>, Mehmet Güzel<sup>1</sup>, Zeynep Dilan Orhan<sup>1</sup>

Van Yuzuncu Yil University, Faculty of Dentistry, Department of Oral and Maxillofacial Surgery, Van,

#### TURKEY

Corresponding author: Levent Ciğerim

Address: Van Yüzüncü Yıl University, Faculty of Dentistry, Department of Oral and Maxillofacial Surgery,

Van, Turkey Postal Code: 65080

E-mail address: levent139@hotmail.com Phone:+905321633287 Office Phone: 904322251744 Fax:

+904322251747

### Levent CİĞERİM

Van Yuzuncu Yil University, Faculty of Dentistry, Department of Oral and Maxillofacial Surgery levent139@hotmailmail.com,
+905321633287, https://orcid.org/0000-0001-5218-8568

### Mehmet GÜZEL

Van Yuzuncu Yil University, Faculty of Dentistry, Department of Oral and Maxillofacial Surgery <a href="mailto:dtmehmetguzel@gmail.com">dtmehmetguzel@gmail.com</a>, +905363609854, <a href="https://orcid.org/0000-0002-9621-0496">https://orcid.org/0000-0002-9621-0496</a>

### Zeynep Dilan Orhan

Van Yuzuncu Yil University, Faculty of Dentistry, Department of Oral and Maxillofacial Surgery <a href="mailto:zeynepdilanorhan@gmail.com">zeynepdilanorhan@gmail.com</a>, +905425525525, <a href="https://orcid.org/0000-0003-1333-9073">https://orcid.org/0000-0003-1333-9073</a>

## VAN YÜZÜNCÜ YIL UNIVERSITY DURSUN ODABAŞ MEDICAL CENTER INFORMED CONSENT FORM FOR RESEARCH

### Dear patient,

Please read this document carefully and listen carefully to what we have said. Detailed information about the research; Detailed information about your rights, benefits and risks of the research can be found in this document. The purpose of these statements is to inform you about your health. Please indicate what you do not understand, your questions will be explained in detail. You can leave the research at any stage of the research if you think that your questions are not adequately explained after you accept to participate in the research or for any other reason. During the research period, the health problems arising from our research will be treated in our hospital immediately. You will not be charged an additional fee for participating in this research, nor will you be paid. Thank you for participating in our research.

### Name of the research:

Evaluation of the Efficacy of Different Drugs in the Treatment of Pain in Patients with Temporomandibular Disorder

### The subject, purpose, method, time and process to be used of the research:

Our research is about temporomandibular joint disorders. Evaluation of different pain relievers in the treatment of pain in Temporomandibular Joint Disorders.

The aim of the study is to evaluate the efficacy of Dexketoprofen Trometamol + Thiocolchicoside, dexketoprofen trometamol + paracetamol and Dexketoprofen Trometamol in the treatment of pain in temporomandibular joint disorders.

### Suggested action/process for research:

The study is planned as randomized, double-blind and prospective. A total of 4 groups of 200 patients, 50 patients in each group, will be included in the study.

Inclusion criteria for the study are as follows: Individuals over 18 years of age, without systemic disease, individuals with pain associated with temporomandibular joint discomfort, individuals who have not undergone interventional procedures related to the temporomandibular joint, individuals who have not used any medication in the last week, individuals without tooth deficiency, in temporomandibular joint imaging individuals with normal findings. Individuals who are allergic to the drugs to be used in the study, pregnant and lactating individuals, and individuals who do not regularly come to the controls will be excluded from the study.

The information of the patients will be recorded in the mother's disease form and the drug to be used will be determined randomly. Patients will use the study drugs regularly for two weeks, and in the following weeks, paracetemol group painkillers will be used if needed. An occlusal plate will be used throughout the entire treatment. During the baseline and control sessions, patients' network levels and other findings will be evaluated. At the end of the 3-month follow-up period, the treatment of patients who need additional treatment will be continued.

Data were collected and evaluated statistically.

Study-specific risks during the study: Allergic reaction

**Possible benefits of the research:** "Dexketoprofen Trometamol + Thiocolchicoside", "Dexketoprofen Trometamol + Paracetomol" and "Dexketoprofen Trometamol" will help to determine the effective drug in the treatment of pain in Temporomandibular Joint Disorders by comparing the pain relief activities.

Dear patient/ participant/....., please read the following articles carefully and fill in the relevant blank or tick the relevant box

| Name surname: Date of birth: Adress: | Associate Professor Levent CİĞERİM<br>Institution Registration Number: 5086<br>Signature: |
|---|---|
| Phone. No: | Name-Surname of the Physician Responsible for the Research: |
| History:: | |
| he Participant's and/or Legal Representative to Get Consent in Emergency Situations | |
| 7. I have the right to withdraw from the research at any time, i know i don't know 8. I will not charge/pay any fee as a result of the research; i know i don't know 9. If a medical risk arises, free medical treatment will be provided. i know i don't know 10. The possible benefits of the research result in detail. i know i don't know 12. When I encounter a health problem during the research; at any hour, Dt. I know that I can call Mehmet GÜZEL at 05363609854 (mobile) and at YYU Faculty of Dentistry, Department of Oral, Dental and Maxillofacial Surgery. | |
| 6. The data received by me regarding the research will be l | kept confidential, i know i don't know |
| treatments, and the procedures to be done. I agree. 5. Since I can't read/write the research information proceduresjoined. | lo not accept. |
| 3. Provided that my identity is kept confidential and used of I may be photographed during the intervention/treatment to retrospectively or recorded. I allow I do not allow. 4. I learned the benefits and possible risks of diagnostic to the confidence of the confi | be applied to me, that my data can be used |
| I agreed. I did not accept. 2. I have read and listened to the points to be considered in the research. I asked my questions about the research. Required enlightening answers I got it, I got it. I didn't get it, I don't understand. | |
| 1. I was invited to the research after I received the prexplained in a clear and simple way and after reading the co | |